CLINICAL TRIAL: NCT07324967
Title: A Standardized Counseling Approach to Preoperative Education in Transmasculine Individuals Receiving Gender-affirming Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OBGYN-2025-34532
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hysterectomy; Gender Affirming Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survey Group (No Intervention)
- Educational Handout + Survey Group (Active Comparator)
  Interventions: Other: Educational Handout

INTERVENTIONS:
Other: Educational Handout — educational handout provided to a randomized cohort of patients that reviews the benefits and risks of retaining ovaries vs removing them. This educational handout will be provided prior to the surgical consultation at the time of the initial survey.
  Arms: Educational Handout + Survey Group

SUMMARY:
The intervention will be an educational handout provided to a randomized cohort of patients that reviews the benefits and risks of retaining ovaries vs removing them. This educational handout will be provided prior to the surgical consultation at the time of the initial survey.

ELIGIBILITY:
Inclusion Criteria:

* Any transgender or non-binary individual
* Age 18-65
* Assigned female at birth who desires a gender-affirming hysterectomy with or without oophorectomy
* English-speaking

Exclusion Criteria:

* Non-transgender individuals
* Any transgender individual who has already had a bilateral oophorectomy
* Any transgender person who was born without ovaries or a uterus
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Score | Day 1
  Lower score = less conflict

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Wise, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States